CLINICAL TRIAL: NCT01249872
Title: Postoperative Thoracic Epidural Analgesia in Super Obese Patients (~BMI 60 kg m-2) Undergoing Open Weight Loss Surgery :Does the Addition of Morphine to 0.1% and 0.2% Levobupivacaine Affect Postoperative Pain Relief, Perioperative Lung Function, Return of Normal Gastrointestinal Mobility and Ambulation?
Brief Title: Patients-Controlled Epidural Analgesia After Gastric Bypass for Morbid Obesity Using Morphine-Levobupivacaine Regimens
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Zotou Natassa,MD, Anesthesiologist M.D, D.E.S.A., University of Patras
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: morbid obesity_post-op pain
Record Dates: First submitted 2010-11-22; First posted 2010-11-30 (Estimated); Results first posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-06

CONDITIONS: Morbid Obesity; Postoperative Pain; Postoperative Bowel Function; Postoperative Ambulation
Keywords: open gastric by-pass; super morbidly obese patients; postoperative thoracic epidural analgesia; different drug regimens (morphine and levobupivacaine); Lung function tests; Postoperative Bowel recovery; Postoperative Ambulation
MeSH Terms: conditions — Obesity, Morbid; Pain, Postoperative | interventions — Morphine; Levobupivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE (Active Comparator): Group A patients receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose 2 ml of normal saline. Postoperatively, patients receive PCEA of 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
  Interventions: Drug: GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE
- GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE (Active Comparator): Group B patients receive an epidural bolus dose of 1mg of morphine intra-operatively (45 min before the estimated end of the surgery). Postoperatively, patients receive PCEA of 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h
  Interventions: Drug: GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE
- GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE (Active Comparator): Group C patients receive an epidural bolus dose 2 mg of morphine intra-operatively (45 min before the estimated end of the surgery).Postoperatively, patients receive PCEA of 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h
  Interventions: Drug: GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE
- GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE (Active Comparator): Group D patients receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 2 ml of normal saline, epidurally. Postoperatively,patients receive PCEA of 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h
  Interventions: Drug: GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE
- GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE (Active Comparator): Group E patients receive intra-operatively (45 min before the estimated end of the surgery) an epidural bolus dose of 1mg of morphine.Postoperatively, patients receive PCEA of 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h
  Interventions: Drug: GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE
- GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE (Active Comparator): Group F patients receive intra-operatively (45 min before the estimated end of the surgery) an epidural bolus dose of 2 mg of morphine. Postoperatively, patients receive PCEA of 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h
  Interventions: Drug: GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE

INTERVENTIONS:
Drug: GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE — Patients receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose 2 ml of normal saline, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA) of 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
  Other Names: Morfina cloridrato 10 mg /ml - Morphine; Chirocaine 5 mg/ml - Levobupivacaine
  Arms: GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE
Drug: GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE — Patients receive intraoperatively(45 min before the estimated end of the surgery)an epidural bolus dose of 1mg of morphine.Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA) of 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
  Other Names: Morfina cloridrato 10 mg /ml - Morphine; Chirocaine 5 mg/ml - Levobupivacaine
  Arms: GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE
Drug: GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE — Patients receive intraoperatively (45 min before the estimated end of the surgery) a bolus dose 2 mg of morphine, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA) of 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
  Other Names: Morfina cloridrato 10 mg /ml - Morphine; Chirocaine 5 mg/ml - Levobupivacaine
  Arms: GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE
Drug: GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE — Patients receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 2 ml of normal saline epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA) of 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
  Other Names: Morfina cloridrato 10 mg /ml - Morphine; Chirocaine 5 mg/ml - Levobupivacaine
  Arms: GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE
Drug: GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE — Patients receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 1mg of morphine, epidurally.Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA) of 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
  Other Names: Morfina cloridrato 10 mg /ml - Morphine; Chirocaine 5 mg/ml - Levobupivacaine
  Arms: GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE
Drug: GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE — Patients receive an epidural bolus dose of 2 mg of morphine intra-operatively (45 min before the estimated end of the surgery).Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA) of 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
  Other Names: Morfina cloridrato 10 mg /ml - Morphine; Chirocaine 5 mg/ml - Levobupivacaine
  Arms: GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE

SUMMARY:
Adequate postoperative analgesia can facilitate recovery following gastric bypass surgery for morbid obesity. The efficacy and safety of intravenous patient - controlled analgesia has been studied, but up to date no data are available concerning the use of thoracic epidural patient-controlled analgesia regarding the use of levobupivacaine combined with morphine in morbidly obese patients. The investigators' aim in this prospective, randomized, double-blinded study was to compare the analgesic effectiveness, the dose requirements and side effects of thoracic epidural patient controlled analgesia 0.1% and 0.2% levobupivacaine combined with a continuous epidural administration of morphine, with or without a loading dose, after open gastric bypass for morbid obesity.

DETAILED DESCRIPTION:
Morbidly obese patients (BMI > 50 kg/m2) planned to undergo open variant of biliopancreatic diversion with Roux-en-Y gastric bypass (BPD-RYGBP) received standardized general anesthesia (intravenous propofol combined with remifentanyl and muscle relaxation). Preoperatively, in all patients an epidural catheter in the thoracic spine level will be placed between T5 and T8 interspace. All patients will be randomly allocated to six groups:

Group A patients will receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose 2 ml of normal saline, epidurally. Postoperatively, immediately after extubation patient controlled epidural anesthesia (PCEA)with 0.1% levobupivacaine (5ml, lockout interval 10min) , combined with a continuous epidural infusion of morphine 0.2 mg/h will be administered, Group B patients will receive an epidural bolus dose of 1mg of morphine intra-operatively (45 min before the estimated end of the surgery) and postoperatively the same levobupivacaine and morphine regimen as Group A, Group C patients will receive an epidural bolus dose 2 mg of morphine intra-operatively and thereafter the same levobupivacaine and morphine regimen as Group A.

Group D patients will receive intra-operatively an epidural bolus dose of 2 ml of normal saline. Postoperatively, the patients will receive PCEA in a dose of 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h, Group E patients will receive intra-operatively an epidural bolus dose of 1mg of morphine intra-operatively and postoperatively the same regimen as Group D.

Group F patients will receive intra-operatively an epidural bolus dose of 2 mg of morphine intra-operatively and thereafter the same regimen as Group D.

Pain assessment will be performed using visual analogue scale (VAS, 10cm scale) at rest, at mobilization and at cough. Furthermore, total local anesthetic and morphine consumption, side effects on cardiovascular, respiratory and gastrointestinal systems, including blood pressure,blood gases, spirometric values Forced Expiratory Volume at 1 sec (FEV1), Forced Vital Capacity (FVC), Peak Expiratory Flow Rate (PEFR), incidents of postoperative nausea and vomiting (PONV), pruritus, time to first flatus, postoperative ambulation will be recorded for up to 6 days.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) > 50
* Age < 50
* Patients written consent to participate in the study

Exclusion Criteria:

* Cardiovascular disease (valvular and ischemic heart disease)
* Patients refusal to participate in the study
* Contraindication to epidural catheter placement (e.g anticoagulation, anti- platelets medication)
* Active psychiatric disease requiring treatment
* Redo surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: KRITON S FILOS, MD, PhD, PROFESSOR, Study Chair — Department of Anesthesiology and Critical Care; ATHINA SIAMPALIOTH, MD, Study Director — University Hospital of Patras; ANASTASIA ZOTOU, MD, Principal Investigator — University Hospital of Patras
Locations (1):
- University of Patras, Department of Anesthesiology and Critical Care Medicine, Pátrai, Achaia, Greece

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2010 and September 2012, a total of 107 morbidly obese patients undergoing an open weight loss surgery (BPD-RYGBP) were assessed for eligibility, with 96 patients randomized to one of the six Groups (n=16)
Pre-assignment Details: From the 107 patients, assessed for eligibility, 11 patients were excluded due to:
  * Surgery postponed (n=3)
  * Decline to participate (n=2)
  * Prolonged surgery >4h, due to complications (n=3)
  * Failure to place epidural catheter (n=3)
Groups:
- GROUP A : 0 mg MORPHINE- 0.1% LEVOBUPIVACAINE: Group A patients (n=16) receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 2ml of normal saline, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP B : 1 mg MORPHINE- 0.1%LEVOBUPIVACAINE: Group B patients (n=16)receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 1mg of morphine, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP C : 2 mg MORPHINE- 0.1% LEVOBUPIVACAINE: Group C patients (n=16) receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 2mg of morphine, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE: Group D patients (n=16)receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 2ml of normal saline, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE: Group E patients (n=16)receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 1mg of morphine, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE: Group F patients (n=16) receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 2mg of morphine, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
Period: Overall Study
Arm/Group | GROUP A : 0 mg MORPHINE- 0.1% LEVOBUPIVACAINE | GROUP B : 1 mg MORPHINE- 0.1%LEVOBUPIVACAINE | GROUP C : 2 mg MORPHINE- 0.1% LEVOBUPIVACAINE | GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE | GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE | GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE
Started | 16 | 16 | 16 | 16 | 16 | 16
Completed | 16 | 16 | 16 | 16 | 16 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE: Group A patients (n=16) receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose 2 ml of normal saline, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE: Group B patients (n=16) receive intraoperatively(45 min before the estimated end of the surgery) an epidural bolus dose of 1mg of morphine.Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE: Group C patients (n=16) receive intraoperatively (45 min before the estimated end of the surgery) an epidural bolus dose 2 mg of morphine. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE: Group D patients (n=16) receive intra-operatively (45 min before the estimated end of the surgery) an epidural bolus dose of 2 ml of normal saline. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE: Group E patients (n=16) receive intra-operatively(45 min before the estimated end of the surgery) an epidural bolus dose of 1mg of morphine. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE: Group F patients (n=16) receive an epidural bolus dose of 2 mg of morphine intra-operatively (45 min before the estimated end of the surgery).Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- Total: Total of all reporting groups
Arm/Group | GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE | GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE | GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE | GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE | Total
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 16 | 16 | 16 | 16 | 96
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years]
  Age (yr) | 35.1 (9.4) | 32.8 (9.5) | 34.8 (9.2) | 34.3 (8.4) | 35.8 (8.1) | 35.1 (8.5) | 34.7 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 12 | 10 | 12 | 9 | 65
  Male | 6 | 4 | 4 | 6 | 4 | 7 | 31
Region of Enrollment [Number; unit: participants]
  Greece | 16 | 16 | 16 | 16 | 16 | 16 | 96
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 57.8 (5.6) | 57.5 (6.0) | 58.3 (7.8) | 58.6 (6.9) | 60.0 (3.9) | 59.4 (7.0) | 58.6 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Scores (Visual Analogue Scale)
Description: Pain scores at rest and on cough using a 10cm Visual Analogue Scale(0=no pain, 10=worst possible pain) were assessed up to 48h postoperatively.
Time Frame: up to 48 h postoperatively
Population: The sample size was chosen in order to detect a difference in the epidural levobupivacaine PCEA consumption at 48 hrs. We calculated that 14 patients per group would be adequate to detect statistical significance (α = 0.05, power = 90%), using data from a previous pilot study Then, we increased the sample size by 15%.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE: Group B patients (n=16) receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 1mg of morphine, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE: Group C patients (n=16)receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 2mg of morphine, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE: Group D patients (n=16)receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose 2 ml of normal saline, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE: Group E patients (n=16) receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 1mg of morphine, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
Arm/Group | GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE | GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE | GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE | GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
units on a scale
  VAS rest at 6h postoperatively | 1.4 (2.3) | 1.6 (1.8) | 1.6 (2.0) | 0.8 (1.4) | 1.1 (1.6) | 0.8 (1.2)
  VAS rest at 24h postoperatively | 0.1 (0.3) | 0.4 (0.9) | 0.4 (1.0) | 0.0 (0.0) | 1.8 (2.0) | 0.1 (0.5)
  VAS rest at 48h postoperatively | 0.0 (0.0) | 0.1 (0.3) | 0.4 (0.9) | 0.0 (0.0) | 0.1 (0.3) | 0.0 (0.0)
  VAS cough at 6h postoperatively | 4.7 (2.7) | 4.2 (2.0) | 4.7 (2.7) | 3.9 (1.9) | 3.9 (1.9) | 2.7 (2.2)
  VAS cough at 24h postoperatively | 2.4 (1.9) | 2.6 (1.9) | 3.2 (2.2) | 2.0 (1.8) | 3.5 (2.0) | 2.4 (1.9)
  VAS cough at 48h postoperatively | 1.3 (1.5) | 2.4 (1.7) | 2.3 (2.3) | 1.3 (1.4) | 1.4 (1.8) | 0.8 (1.2)

2. Secondary Outcome: Time to Postoperative Bowel Recovery
Description: Time to postoperative recovery of bowel function assessed by first flatus or stool, noticed by the patient
Time Frame: up to 6 days
Measure: Mean (Standard Deviation); unit: hours
Groups:
- GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE: Group A patients (n=16) receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 2ml of normal saline, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE: Group C patients (n=16) receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 2mg of morphine, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
- GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE: Group D patients (n=16) receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 2ml of normal saline, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
Arm/Group | GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP B : 1 mg MORPHINE- 0.1%LEVOBUPIVACAINE | GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE | GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE | GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
hours | 56.6 (11.9) | 70.9 (11.9) | 67.1 (11.8) | 55.6 (12.7) | 58.6 (14.5) | 63.9 (12.0)

3. Secondary Outcome: Time to First Postoperative Ambulation
Description: Time to being able to walk without assistance within the room or outside the room
Time Frame: up to 6 days
Measure: Mean (Standard Deviation); unit: hours
Groups:
- GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE: Group B patients (n=16)receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 1mg of morphine, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.1% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
Arm/Group | GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE | GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE | GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE | GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
hours
  Walking in the room unassisted | 19.0 (4.1) | 19.9 (3.4) | 19.1 (3.5) | 20.7 (4.6) | 21.4 (1.9) | 20.6 (3.3)
  Walking out of the room unassisted | 33.3 (12.1) | 47.0 (11.1) | 43.3 (11.1) | 39.5 (14.0) | 43.4 (11.6) | 45.1 (10.7)

4. Secondary Outcome: Consumption of Levobupivacaine at 24h and 48 h Postoperatively
Description: Cumulative consumption of levobupivacaine administered via patients controlled epidural analgesia pump( PCEA) at 24h and 48 h postoperatively
Time Frame: up to 48 hours postoperatively
Measure: Mean (Standard Deviation); unit: mg
Groups:
- GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE: Group F patients (n=16)receive intra-operatively (45 min before the estimated end of the surgery) a bolus dose of 2mg of morphine, epidurally. Postoperatively, immediately after extubation, patients receive patient controlled epidural analgesia (PCEA)with 0.2% levobupivacaine (5ml, lockout interval 10min) combined with a continuous epidural infusion of morphine 0.2 mg/h.
Arm/Group | GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE | GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE | GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE | GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
mg
  Levobupivacaine consumption at 24h postoperatively | 132.9 (58.9) | 178.8 (90.1) | 165.6 (92.9) | 325.7 (147.2) | 241.9 (145.0) | 203.1 (115.2)
  Levobupivacaine consumption at 48h postoperatively | 189.8 (117.5) | 240.9 (133.0) | 231.9 (139.2) | 435.4 (220.2) | 351.3 (193.6) | 294.7 (158.0)

5. Secondary Outcome: Cumulative Consumption of Epidural Morphine at 24h and 48h Postoperatively
Description: Cumulative consumption of epidural morphine administered as loading dose, intraoperatively, of 1mg(groups B and E)or 2mg (groups C and F) and as continuous infusion of 0,2mg/h ( all groups) at 24h and 48h postoperatively.All participants in each Group received the same dose of epidural morphine, as no participant missed a scheduled dose.
Time Frame: up to 48 hours postoperatively
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE | GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE | GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE | GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
mg
  Epidural morphine consumption at 24h postoperative | 4.8 (0.0) | 5.8 (0.0) | 6.8 (0.0) | 4.8 (0.0) | 5.8 (0.0) | 6.8 (0.0)
  Epidural morphine consumption at 48h postoperative | 9.6 (0.0) | 10.6 (0.0) | 11.6 (0.0) | 9.6 (0.0) | 10.6 (0.0) | 11.6 (0.0)

6. Secondary Outcome: Change From Baseline of Spirometric Values
Description: Preoperatively, after a detailed demonstration, baseline spirometry measurements of forced vital capacity (FVC), forced expiratory volume in 1 s (FEV1) and peak expiratory flow rate (PEFR) were measured, using a bedside spirometer (PowerCubeΤΜ, Ganshorn Medizin Electronic, Germany), on-line connected to a PC. Spirometry was standardized with each patient in a 30o head-up position and it was performed at least three times and the best measurement was recorded, according to the criteria of the European Respiratory Society .Postoperatively, spirometric values (FVC= Forced Vital Capacity, FEV1=Forced Expiratory Volume at 1 sec , PEFR= Peak Expiratory Flow Rate)were recorded at 12, 24, 36, 48, 72, 144 hours . Data are expressed as percentage of preoperative values, which are 100%.
Time Frame: up to 6th day postoperatively
Measure: Mean (Standard Deviation); unit: percentage of preoperative values
Arm/Group | GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE | GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE | GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE | GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
percentage of preoperative values
  FVC at 12h postoperatively | 63.2 (15.2) | 69.3 (13.1) | 68.3 (15.9) | 71.7 (14.0) | 66.4 (11.3) | 66.8 (14.6)
  FVC at 24h postoperatively | 62.5 (15.6) | 62.2 (13.7) | 72.1 (15.5) | 66.8 (15.6) | 63.3 (12.1) | 62.6 (12.3)
  FVC at 36h postoperatively | 65.7 (13.6) | 61.2 (13.8) | 65.2 (15.5) | 63.9 (13.4) | 62.8 (14.6) | 63.2 (9.3)
  FVC at 48h postoperatively | 63.9 (15.0) | 66.2 (12.5) | 67.6 (13.4) | 69.8 (10.1) | 71.1 (15.0) | 66.9 (10.9)
  FVC at 72h postoperatively | 69.4 (7.0) | 71.3 (11.8) | 76.2 (16.8) | 72.4 (10.9) | 77.3 (15.1) | 76.7 (9.0)
  FVC at 6th day postoperatively | 79.0 (18.3) | 83.9 (7.6) | 83.1 (8.0) | 84.0 (11.5) | 80.0 (18.2) | 89.2 (9.6)
  FEV1 at 12h postoperatively | 55.8 (19.3) | 63.9 (11.7) | 60.5 (15.3) | 65.2 (15.1) | 62.0 (9.3) | 62.1 (18.6)
  FEV1 at 24h postoperatively | 61.5 (17.1) | 55.2 (18.4) | 71.0 (15.0) | 63.8 (16.4) | 56.4 (14.8) | 59.8 (12.1)
  FEV1 at 36h postoperatively | 62.9 (15.4) | 52.7 (16.4) | 61.0 (16.2) | 58.4 (14.2) | 61.1 (16.3) | 59.3 (11.4)
  FEV1 at 48h postoperatively | 64.9 (18.1) | 55.9 (22.5) | 68.2 (19.6) | 61.8 (8.8) | 67.1 (12.6) | 64.9 (11.6)
  FEV1 at 72h postoperatively | 79.0 (26.1) | 70.2 (15.0) | 75.4 (8.5) | 70.2 (15.0) | 75.3 (8.5) | 72.5 (10.0)
  FEV1 at 6th day postoperatively | 86.8 (23.5) | 81.8 (7.9) | 88.0 (12.9) | 83.4 (12.0) | 79.4 (15.9) | 83.8 (8.7)
  PEFR at 12h postoperatively | 62.9 (32.3) | 67.6 (21.1) | 61.8 (20.9) | 60.0 (22.8) | 77.9 (22.6) | 67.2 (25.6)
  PEFR at 24h postoperatively | 68.5 (21.8) | 55.6 (21.3) | 79.9 (14.3) | 70.1 (13.6) | 57.7 (22.0) | 68.9 (12.8)
  PEFR at 36h postoperatively | 69.6 (22.0) | 57.9 (27.8) | 68.8 (20.6) | 59.4 (18.0) | 73.8 (25.6) | 67.9 (20.3)
  PEFR at 48h postoperatively | 70.7 (27.4) | 58.8 (29.2) | 79.7 (25.8) | 64.9 (17.7) | 76.4 (23.6) | 74.3 (11.8)
  PEFR at 72h postoperatively | 77.3 (26.5) | 78.1 (32.0) | 91.3 (35.0) | 70.7 (15.1) | 80.9 (19.3) | 86.0 (28.8)
  PEFR at 6th day postoperatively | 93.8 (31.5) | 98.4 (34.6) | 96.4 (15.3) | 76.3 (16.1) | 83.7 (20.5) | 89.6 (19.5)

ADVERSE EVENTS:
Time Frame: Adverse effects (opioid or epidural related) were assessed during the in hospital postoperative period (6days)
Description: Clinical observation and reported by the patient
Arm/Group | GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE | GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE | GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE | GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE | GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE
Serious Adverse Events (participants affected / at risk) | 0/16 | 3/16 | 3/16 | 0/16 | 2/16 | 3/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GROUP A : 0 mg MORPHINE-0.1% LEVOBUPIVACAINE (N=16) | GROUP B : 1 mg MORPHINE- 0.1% LEVOBUPIVACAINE (N=16) | GROUP C : 2 mg MORPHINE-0.1% LEVOBUPIVACAINE (N=16) | GROUP D : 0 mg MORPHINE- 0.2% LEVOBUPIVACAINE (N=16) | GROUP E : 1 mg MORPHINE-0.2 % LEVOBUPIVACAINE (N=16) | GROUP F : 2 mg MORPHINE- 0.2% LEVOBUPIVACAINE (N=16)
Postoperative nausia and vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
Postoperative pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
* Patients in groups A and D did not receive epidural morphine intraoperatively.
* We excluded patients aged > 50 yr as increasing the age of morbidly obese patients, might have increased the risk of perioperative complications

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes